CLINICAL TRIAL: NCT02635321
Title: MRI and Muscle Involvement in Patients With Mutations in GMPPB
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sofie Thurø Østergaard, Bachelor of Science, Rigshospitalet, Denmark
Other Study IDs: STO-GMPPB
Record Dates: First submitted 2015-12-01; First posted 2015-12-18 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Limb-girdle Muscular Dystrophy
Keywords: MRI; LGMD; GMPPB
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with LGMD 2T: Four patients over 18 years old with genetically verified LGMD 2T.

SUMMARY:
Limb girdle muscular dystrophies (LGMD) are a very heterogeneous group of muscle disorders characterized by muscle weakness and atrophy of the proximal muscles of the shoulder and pelvic girdles. LGMD is classified based on its inheritance pattern and genetic cause into more than 31 different types.

A new type - type 2T has been found. The genetic cause of type 2T is mutations in Guanosine Diphosphate (GDP)-mannose pyrophosphorylase B (GMPPB). Mutations in GMPPB can also cause Congenital muscular dystrophies (CMD). Only 41 patients with mutations in GMPPB has been reported.

In this study, the investigators examine five new cases with the LGMD phenotype. The primary aim is to examine the muscle involvement using MRI.

ELIGIBILITY:
Inclusion Criteria:

* Persons with genetically verified mutations in GMPPB

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons diagnosed with mutations in GMPPB in Denmark and France are invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
MRI scan for qualitative analysis of muscle involvement | One MRI scan per subject (exam lasts approximately 60 min.)
  The MRI protocol include T1-weighted brain and whole body examination. Four cross-sectional slices at shoulder, lumbar back, thigh and calf are chosen for qualitative analysis using the grading scale developed by Mercuri et al. (2007).

SECONDARY OUTCOMES:
Muscle biopsy for biochemical investigation | One muscle biopsy per subject (last approximately 15 min.)
  Muscle biopsies from the tibialis anterior muscle and the deltoid muscle will be analyzed for glycosylated α-dystroglycan, merosin and GMPPB. (Concentration determined by standard biochemical analysis).
10 meter walk test | Exam last approximately 5 min.
  Measurement of the time it takes to walk 10 meters.
Neurological examination and test of muscle strength | Exam last approximately 15 min.
  Muscle strength (in arms and legs) will be examined based on the Medical Research Council (MRC) scale.
Questionnaires | Data will be collected once for patients with LGMD 2T (exam last approximately 45 min.)
  Data will be collected using Minimal mental examination (MMSE) and Fatigue Severity Scale (FSS).
Heart examination | Exam last approximately 45 min
  Echocardiography and Electrocardiogram (ECG).
Forced Vital Capacity (FVC) | Exam last approximately 15 min
  FVC is measured as the best of three attempts using a hand-held spirometer.
Electromyography (EMG) | Exam last approximately 30 min
  EMG is used for measuring nerve conducting velocity and neuromuscular activity.

CONTACTS AND LOCATIONS:
Overall Officials: Sofie T Østergaard, Bsc., Principal Investigator — Copenhagen Neuromuscular Center, Department of Neurology, Rigshospitalet, Copenhagen University
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Copenhagen, Denmark